CLINICAL TRIAL: NCT03345563
Title: Biobehavioral Effects of Tai Chi Qigong (TCQ) for Male Cancer Survivors With Fatigue (HERO)
Brief Title: Project HERO: Health Empowerment & Recovery Outcomes
Acronym: HERO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: University of California, Los Angeles (Other); University of New Mexico (Other)
Responsible Party: Principal Investigator, Anita Y. Kinney, PhD, RN, Study Principal Investigator; Associate Director for Cancer Health Equity, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 131816; Pro2018002020 (Other: Rutgers, The State University of New Jersey)
Record Dates: First submitted 2017-11-06; First posted 2017-11-17 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer; Bladder Cancer; Kidney Cancer; Colon Cancer; Rectum Cancer; Thyroid Cancer; Lung Cancer; Small Intestine Cancer; Soft Tissue Cancer
Keywords: Prostate Cancer; Fatigue; Elderly; Supportive Care; Light Exercise; Quality of Life; Bladder Cancer; Kidney Cancer; Colon Cancer; Rectum Cancer; Throid Cancer; Lung Cancer; Small Intestine Cancer; Soft Tissue Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Bladder Neoplasms; Kidney Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Thyroid Neoplasms; Lung Neoplasms; Sarcoma; Fatigue

STUDY DESIGN:
Intervention Model Description: After obtaining informed consent and baseline assessments, cancer survivors aged 55 years and older with some level of fatigue will be randomized to the BMT arm or intensity-matched Body Training (BT), or Usual Care (UC) arms. Patient-reported assessments (surveys) will occur at baseline (within 2-weeks pre- intervention), mid-intervention (6 weeks), 1-week post-intervention (13 weeks), and at 3 months and 12 months post-intervention. Phlebotomy is done at baseline, 1 week post intervention (13 weeks), and 3 months and 12 months post intervention. Dietary assessments are done at baseline, and week 13 (1 week post intervention), 3 months and 1 year post-intervention. Physical activity is assessed weekly throughout the intervention. Sleep diaries are collected at all time points.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Participants will be instructed not to discuss their arm assignment with study personnel during their assessments. We avoided the use of the terms Tai Chi and Qigong for participant recruitment, patient-faced materials, and intervention implementation. Questionnaires will be self-administered, administered in person or by telephone based on participant need and preference. Some investigators, the data manager, biostatisticians, biometric testing and lab technicians will be blinded to intervention allocation. The technicians who analyze biospecimens will be blinded to all other data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Body Mind Training (BMT) (Experimental): Body mind training
  Interventions: Behavioral: Body Mind Training (BMT)
- Body Training (BT) (Active Comparator): Body training only
  Interventions: Behavioral: Body Training (BT):
- Usual care (UC): (Other): Control
  Interventions: Behavioral: Usual Care (UC)

INTERVENTIONS:
Behavioral: Body Mind Training (BMT) — Participants will practice BMT under the instruction of a BMT instructor. There will be 24 sessions. Each session will last 60 minutes and will occur twice a week for 12 weeks. Each session will include both light physical exercise and mind training.
  Sessions will be supplemented with home-based practice using an instructional DVD and handouts. Participants will be instructed to practice at least 30 minutes a day (at least 3 days per week) throughout the intervention and post-intervention period.
  Arms: Body Mind Training (BMT)
Behavioral: Body Training (BT): — Participants will practice BT under the instruction of a BT instructor. There will be 24 sessions. Each session will last 60 minutes and will occur twice a week for 12 weeks. Sessions will be supplemented with home-based practice using an instructional DVD and handouts. Participants will be instructed to practice at least 30 minutes a day (at least 3 days per week) throughout the intervention and post-intervention period.
  Arms: Body Training (BT)
Behavioral: Usual Care (UC) — Participants in the usual care arm will receive care as normal and will not attend classes but will complete the same assessments as participants in the BMT and BT classes.
  Arms: Usual care (UC):

SUMMARY:
Project HERO is a 12-week study of the efficacy of Body Mind Training (BMT, i.e. Tai Chi and Qigong in this project) for reducing fatigue in male cancer survivors. This 3-arm randomized clinical trial will examine inflammatory biology and selected gene-expression pathways that are hypothesized to contribute to the intervention's effect.

DETAILED DESCRIPTION:
This study will establish the efficacy of a 12-week Body Mind Training (BMT) for reductions in fatigue (the study's primary outcome). Secondary patient-reported outcomes include quality of life changes (e.g., changes in sleep and perceived psychological distress), changes in the biomarkers of inflammation, including genome-wide transcriptional factors, and expression of fatigue-related genes. Post-award, the target sample size was revised to (n=166) with NCI permission.

There are over 9 million cancer survivors who are 55 years of age or older. Cancer survivors in this age group have unique challenges coping with the late and long-term effects of having had a cancer diagnosis and treatment, coupled with age-related declines and comorbidities. This may influence their ability to engage in lifestyle interventions because of slower post-treatment recovery, increased functional limitations, and other quality of life (QOL) impairments. Fatigue is common, under-recognized, undertreated, and correlated with impairments in psychological distress, social and functional well-being, and health-related QOL in cancer survivors. For male cancer survivors suffering from fatigue, Tai Chi and Qigong (TCQ) may be more appealing because it is not overly physically exertive and is safe for people 55 years of age or older. In this study, we referred to the intervention groups as follows: TCQ intervention was referred to as body-mind training (BMT), and the exercise intensity-matched condition was referred to as body training (BT). This was done to help reduce bias by minimizing participants' expectations or perceived differences between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 55 years
* Previous diagnosis of local, regional, or metastatic cancer. If treated for cancer, prostate cancer therapy completed, 3+ months. If on ADT/ hormone manipulation, must be for 4 or more months
* Previous diagnosis of small intestine, thyroid, oral, non-muscle invasive bladder, kidney/renal, lung, colon, rectum, soft tissue, or other cancer
* Meet study criteria for fatigue: Medical Health Outcome Study Short Form Vitality/Fatigue subscale (SF-36 Vitality scale-4 items; 5 Likert scale) using a fatigue cut-off value of ≤13; or the Patient-Reported Outcomes Measurement Information System Fatigue scale (PROMIS Fatigue scale) using a cut-off value of ≥9
* Live within 75 miles of New Brunswick or Newark
* Inactive (<150 minutes of vigorous exercise/week within the past 3 months)
* Has transportation to attend on-site classes and assessments

Exclusion Criteria:

* Patient Health Questionnaire PHQ-9 Score >12
* Indication of suicidality from PHQ-9 reports that he has several or more days of "thoughts that you would be better off dead, or of hurting yourself."
* Karnofsky performance status score of 50 or below
* Current regular practice within the past year (2-3 times a week over a period of two months that is not interrupted) of BMT or other complementary and alternative medicine that shares similar principles of BMT.
* Inability to speak and read English proficiently
* Unable to understand informed consent
* Current health conditions that may interfere with the intervention: respiratory, cardiovascular, or neurological problems unless released by a physician
* Medical conditions or activities that can cause severe fatigue: Severe hearing loss that would cause difficulty following an instructor in a group setting, chronic fatigue syndrome, current major depression, alcohol use disorder, shift work
* Prostate cancer that has metastasized to the liver, brain, or lungs
* Currently receiving chemotherapy with VePesid, Cytoxan, Enzalutamide (XTANDI®), intravenous chemotherapy or radionucleotides (Strontium-89, Samarium (Quadramet®), Radium-223 (Xofigo®)), or other therapy (as confirmed by study team)
* Unwilling to be randomized to study arms and/or commit to 12 weeks of classes and assessments
* Have had a diagnosis of another cancer, unless:

  * Non-melanoma skin cancer or
  * Completed treatment AND cancer-free for 5 or more years.

We will not include any of the following special populations:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Min Age: 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Functional Assessment of Chronic Illness (FACIT)-Fatigue Scale | Baseline (2 weeks pre-intervention) and week 6, and post-intervention at week 13, 3 months, and 12 months
  Change in fatigue levels from baseline to 3-months post intervention: measured with 13-item scale assessing the level of fatigue during usual activities over the 7 days prior to the measurement timepoint, with higher scores indicating less fatigue. Administered at several time points to measure the effect the intervention.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | Baseline (2 weeks pre-intervention) and week 6, and post-intervention at week 13, 3 months, and 12 months
  Questionnaire: Measures sleep disturbance with 19 items, generating seven component scores: Subjective sleep quality, Sleep latency, Sleep duration, Habitual sleep efficiency, Sleep disturbances, Use of sleeping aid medication(s), and Daytime dysfunction. The global PSQI score is a composite of the 7 component scores, ranging from 0 to 21, which was used in this study.
Inflammation Biology Measures: Changes in circulating levels pro- and anti-inflammatory biomarkers will be assessed by measuring NF-κB and AP-1. | Baseline (2 weeks pre-intervention), and post-intervention at week 13, 3 months, and 12 months
  Blood samples will be collected at using standardized procedures. The dynamics of inflammation will be measured by using a vertically integrated mechanistic approach and examining upstream signaling pathways and circulating levels. Circulating levels will be assessed by assay of plasma pro- and anti-inflammatory biomarkers; Inflammatory signaling as indexed by activation of key inflammatory transcription factors (e.g., NF-κB) will be measured using intranuclear staining and flow cytometric analyses. Genome-wide transcriptional analyses (all baseline and 13-week biospecimens) will be used to identify the differential regulation of gene expression and the molecular inflammation-related signaling pathways that are plausible candidates driving these changes (e.g., NF-κB).
Gene Expression | Baseline (2 weeks pre-intervention), and post-intervention at week 13, 3 months, and 12 months
  Specimen collection and analysis to measure mRNA intercorrelations: 1) Inflammation, Vasodilation, and Metabolite Sensing and 2) Energy and Adrenergic Activation.
Brief Symptom Inventory-18 (BSI-18) | Baseline (2 weeks pre-intervention) and week 6, and post-intervention at week 13, 3 months, and 12 months
  Questionnaire: Psychological distress (depression and anxiety) is measured using the using the Brief Symptom Inventory-18 instrument. Items are summed to calculate the raw score, range 0-72. Raw scores can be converted to T-scores, based on US population norms. Participants with T-scores that are ≥ 63 are considered a "case," and may need professional help. Somatization Scale: Raw score range 0-24, with 24 indicating high somatization. Depression Scale: Raw score range 0-24, with 24 indicating high depression. Anxiety Scale: Raw score range 0-24, with 24 indicating high anxiety.
SF-36v2 Health-Related Quality of Life Survey (Mental and Physical) | Baseline (2 weeks pre-intervention) and week 6, and post-intervention at week 13, 3 months, and 12 months
  Questionnaire: Provides scores for each of the eight health domains and psychometrically-based physical component summary (PCS) and mental component summary (MCS) scores. The raw score of each of the eight SF-36 dimensions was derived by summing the item scores. Subtract the lowest possible raw score from the actual raw score, divide by the possibly raw score range, and multiply by 100 to get the transformed scale. Higher scores indicate better health-related quality of life.
Consensus Sleep Diary | Baseline (2 weeks pre-intervention) and week 6, and post-intervention at week 13, 3 months, and 12 months
  The sleep diary is designed to gather information about daily sleep patterns. Sleep diary is maintained for 7 days prior to each data collection time point.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Y Kinney, PhD, RN, Principal Investigator — Rutgers, The State University of New Jersey; Michael R. Irwin, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Rutgers University, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kinney AY, An J, Lin Y, Tundealao S, Saraiya B, Lu SE, Guest DD, Harding EM, Amorim F, Heidt E, Arana-Chicas E, Chen C, Boyce T, Kim IY, Arap W, Blair CK, Irwin MR. Project HERO: a randomized trial of Tai Chi qigong versus intensity-matched exercise and usual care for fatigue in older male cancer survivors. BMC Complement Med Ther. 2025 Jul 4;25(1):239. doi: 10.1186/s12906-025-04988-7. PMID 40616105

DOCUMENTS (1):
  • Informed Consent Form (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/63/NCT03345563/ICF_000.pdf